CLINICAL TRIAL: NCT05177081
Title: Feasibility of Treatment Using Home Bioelectrical Impedance Analysis and Linked Application System in Patients With Heart Failure: A Multicenter Study
Brief Title: Home BIA Management System in Patients With Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Eung Ju Kim, Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BWA ON Pilot
Record Dates: First submitted 2022-01-03; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Heart Failure，Congestive
Keywords: Heart failure; Bioelectrical impedance analysis
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: multi-center, open label, randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Home BIA Monitoring group (Experimental): Preemptive management by Body fluid monitoring system (BWA ON + App + Web)
  Interventions: Device: Preemptive management using home BIA monitoring system
- Control group (No Intervention): Usual heart failure management (Outpatient follow-up and medical treatment)

INTERVENTIONS:
Device: Preemptive management using home BIA monitoring system — Patients check their body composition and fluid using Home BIA system. Investigators analyze patients' body congestion status and send patient's edema status and direction of extra-diuretics usage to enrolled patients every one week.
  Arms: Home BIA Monitoring group

SUMMARY:
This study is a prospective, multi-center, open label, randomized clinical trial conducted in the republic of Korea. The objective of this study is to evaluate the efficacy and safety of the treatment using home bioelectrical impedance analysis (BIA) and linked application system in patients with heart failure (HF).

DETAILED DESCRIPTION:
The prevalence of HF is generally estimated at 1% to 2% of the general population. The more concerning thing is that HF patients are rapidly increasing due to an increase of elderly population derived from life extension; an increase in the number of survivors of heart disease due to the development of medical technology; and an increase in risk factors for HF such as obesity, diabetes, and ischemic heart disease.

HF is known that a quarter of HF patients are readmitted within 1 year, and the mortality rate within 5 years is about 50%. HF is a chronic condition, punctuated by acute decompensated episodes. Each acute decompensated event results in further organ damage: myocardial and renal damage occurring during such episodes may contribute to progressive left ventricular and/or renal dysfunction. Increasing frequency of acute events with disease progression leads to higher rates of hospitalization and increased risk of mortality.

The main symptoms of HF are shortness of breath and swelling, which are the main reasons for visiting the emergency room and hospitalization. After discharge, body water monitoring and management of HF patients are very important to prevent HF aggravation and re-hospitalization.

There are several methods of body fluid monitoring in HF patients. Current guidelines of heart failure recommends monitoring of pulmonary artery pressures using a wireless implantable hemodynamic monitoring system in symptomatic HF patients with previous HF hospitalization. Multi-parameter monitoring based on ICD is also recommended in order to improve clinical outcomes in HF patients. However, existing HF monitoring and management systems have limitations of its invasiveness, expensive costs and a lot of medical providers' efforts. Other body water monitoring methods are signs and symptoms monitoring and body weight-based monitoring. However, signs such as weight gain and edema or symptoms like dyspnea due to worsening heart failure were not recognized until just 7 and 3 days before the hospitalization event.

BIA, Bioelectrical impedance analysis can be a novel option for body water monitoring method in HF patients. Nowadays, it is possible to obtain more accurate body water by reflecting both intracellular and extracellular water by using multiple frequencies, and it is possible to accurately measure body water even in patients with unusual body water conditions such as heart failure status. Moreover, the changes of Bioelectrical Impedance are detected about two weeks before heart failure hospitalization. It is the key benefit for congestion monitoring and management.

Previous studies have shown that monitoring body water through non-invasive bioelectrical impedance can predict the worsening of HF even in patients with heart failure. In addition, there are studies that reported improvement of clinical results during treatment based on the edema index (extracellular water / total body water) during body water monitoring through non-invasive bioelectrical impedance.

Home BIA monitoring using BWA-ON has potential benefit for continuous water monitoring for edema control in patients with HF. Therefore, we aim to evaluate feasibility of treatment using home BIA and linked application system in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed heart failure
2. Patients taking loop diuretics for HF symptom control
3. Patients who can use a smart-phone

Exclusion Criteria:

1. Patients with implanted devices that could interfere with the BIA such as ICD and CRT
2. Patients with limb defects
3. Patients who unable to stand alone
4. Patients who are pregnant
5. Patients with End-stage renal disease (ESRD) on hemodialysis, serum creatinine of more than 5mg/dL, or nephritic syndrome
6. Patients with systemic diseases such as hypothyroidism, decompensated liver cirrhosis, and systemic lupus erythematosus.
7. Patients with active cellulitis, severe varicose vein, deep vein thrombosis or lymphedema

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in NT-proBNP | 3 months
  NT-proBNP

SECONDARY OUTCOMES:
Rate of heart failure hospitalizations (HHF) | 3 months
  Hospitalization for heart failure
Change from baseline in edema index using BIA | 3 months
  Edema index by BIA
Change from baseline in Creatinine | 3 months
  Creatinine
Change from baseline in symptom of dyspnea | 3 months
  NYHA classification and VAS scale of dyspnea

CONTACTS AND LOCATIONS:
Overall Officials: Eung Ju Kim, MD, PhD, Principal Investigator — Korea University Guro Hospital
Locations (2):
- South Korea (2):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do
  - Korea University Guro Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No